CLINICAL TRIAL: NCT06563739
Title: Director of Rehabilitation Medicine
Brief Title: Study on the Application of Shock Wave Technique After Rotator Cuff Operation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2024520
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Rotator Cuff Tear
Keywords: Shock wave technique
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Exposed group1 (Experimental): Patients who receive divergent low energy once a week
  Interventions: Procedure: Divergent low energy shock wave
- Exposed group2 (Experimental): Patients who receive divergent low energy twice a week
  Interventions: Procedure: Divergent low energy shock wave
- Exposed group3 (Experimental): Patients who recieve divergent medium and low energy once a week
  Interventions: Procedure: Divergent medium and low energy shock wave
- Exposed group4 (Experimental): Patients who receive divergent medium and low energy twice a week
  Interventions: Procedure: Divergent medium and low energy shock wave
- Exposed group 5 (Experimental): Patients who receive focused low energy once a week
  Interventions: Procedure: Focused low energy shock wave
- Exposed group6 (Experimental): Patients who receive divergent medium energy once a week
  Interventions: Procedure: Divergent medium energy shock wave
- Exposed group 7 (Experimental): Patients who receive divergent medium energy twice a week
  Interventions: Procedure: Divergent medium energy shock wave
- Non-exposed group (Experimental): Patients who receive rehabilitation assessment and training guidance
  Interventions: Procedure: Non-exposed group

INTERVENTIONS:
Procedure: Divergent low energy shock wave — Receive divergent low energy shock wave once a week
  Arms: Exposed group1
Procedure: Divergent low energy shock wave — Receive divergent low energy shock wave twice a week
  Arms: Exposed group2
Procedure: Divergent medium and low energy shock wave — Receive divergent medium and low energy shock wave once a week
  Arms: Exposed group3
Procedure: Divergent medium and low energy shock wave — Receive divergent medium and low energy shock wave twice a week
  Arms: Exposed group4
Procedure: Focused low energy shock wave — Receive focused low energy shock wave once a week
  Arms: Exposed group 5
Procedure: Divergent medium energy shock wave — Receive divergent medium energy shock wave once a week
  Arms: Exposed group6
Procedure: Divergent medium energy shock wave — Receive divergent medium energy shock wave twice a week
  Arms: Exposed group 7
Procedure: Non-exposed group — Traditional rehabilitation assessment and training guidance
  Arms: Non-exposed group

SUMMARY:
This study is a prospective cohort study and is a single-center clinical trial. The subjects of this study were patients who underwent rotator cuff repair in the Department of Sports Medicine and the Department of Rehabilitation in the Third Hospital of Beijing Medical University. The sample size of this study is about 2600 cases. We will collect the results of shoulder joint function score, quality of life score, pain score and MRI examination of all participants at baseline. Meanwhile, epidemiological data and related clinical characteristics of patients will be collected at the time of enrollment. All the collected data information was entered into the computer for statistical analysis, and the prognosis of patients under different programs was evaluated.

DETAILED DESCRIPTION:
The shoulder joint is the most flexible joint in the body, and the rotator cuff is an important structure to maintain its stability, and the flexibility of the shoulder joint also leads to joint instability leading to rotator cuff tears, especially in the elderly, previous studies have shown that the incidence of rotator cuff tears in people under the age of 20 is 9.7%, and the incidence of rotator cuff tears in people over the age of 80 can reach 62%. Rotator cuff tears are a common cause of limited mobility and pain in the shoulder joint, severely affecting patients' quality of life. Young people, high-level athletes and sports enthusiasts also have a higher risk of rotator cuff injury.

Arthroscopic rotator cuff repair is widely used in the treatment of rotator cuff tears, and has many advantages such as less postoperative tissue damage, less surgical scar, less infection, and faster recovery. However, its postoperative rehabilitation has always been a hot topic of research. The basic goal of rehabilitation is to protect tendons, promote their healing, prevent shoulder stiffness and muscle atrophy.

In recent years, there have been clinical studies on the application of ESWT in arthroscopic postoperative patients, but its efficacy is still different . However, few clinical studies have been conducted to investigate the effects of ESWT on functional recovery, tendon recovery and MRI imaging after arthroscopic rotator cuff repair. In addition, currently, the application of shock wave technology in the treatment of patients after rotator cuff surgery is very confusing, and there is no clear optimal treatment plan.

In conclusion, the purpose of this study is to compare the difference in efficacy of postoperative rehabilitation programs of different ESWT combined with conventional rehabilitation training on patients after rotator cuff repair, the impact of ESWT on clinical efficacy of patients after rotator cuff repair, and to explore the application of shock wave technology for accurate diagnosis and treatment of rotator cuff surgery

ELIGIBILITY:
Inclusion Criteria:

1. A rotator cuff tear was diagnosed and surgery was required
2. Able to complete cardiopulmonary exercise tests
3. Able to cooperate with rehabilitation training and complete questionnaire survey

Exclusion Criteria：

1. Age <17 years or age >75 years
2. Previous shoulder surgery history
3. Irreparable rotator cuff damage

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
pain VAS score | 6 weeks, 3 months, and 6 months after surgery
  pain levels in patients, ranging from 0 to 10, with a higher score indicating more intense pain.
ASES score | 6 weeks, 3 months, and 6 months after surgery
  The American Shoulder and Elbow Surgeons (ASES) score is the most commonly used score to describe the function of patients' shoulder joints, ranging from 0 to 100. The higher the score, the better the function of patients' shoulder joints.

SECONDARY OUTCOMES:
Active shoulder ranges of motion | 6 weeks, 3 months, and 6 months after surgery
  internal rotation at the side, and external and internal rotation at 90° of abduction

CONTACTS AND LOCATIONS:
Overall Officials: Guoqing Cui, Study Chair — Peking University Third Hospital
Locations (1):
- PekingUTH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No